CLINICAL TRIAL: NCT00781365
Title: Home Blood Pressure Telemonitoring and Case Management to Control Hypertension
Acronym: Hyperlink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07116; 1R01HL090965 (NIH); 2R01HL090965 (NIH)
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Hypertension
Keywords: Hypertension; Telemonitoring; Pharmacy management
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Patients in the control group will receive usual care from their primary care physicians at HealthPartners Medical Group clinics.
- Telemonitors and pharmacy management (Experimental): The telemonitoring intervention (TI) patients will receive a home blood pressure telemonitor and will work with a clinical pharmacist case manager to control elevated blood pressure. Patients will use their home telemonitors to read and send their blood pressures to their Pharmacist case manager, who will use phone meetings with the patient to make medication adjustments.
  Interventions: Other: Telemonitors and pharmacy management

INTERVENTIONS:
Other: Telemonitors and pharmacy management — Patients in the intervention arm will receive home blood pressure monitors, and will have individual hypertension case management from a medication therapy management pharmacist.
  Arms: Telemonitors and pharmacy management

SUMMARY:
In this project we develop and implement an intervention to improve hypertension control in a primary care setting that takes advantage of new technology (home blood pressure telemonitoring) and team models of care (pharmacist case management). The results of the project will have important implications for future efforts to improve care provided to many of the estimated 20 million Americans with uncontrolled hypertension.

DETAILED DESCRIPTION:
Blood pressure (BP) is controlled to recommended levels in only 1 in 3 people with hypertension, and there has been little improvement since the late 1980s, despite advances in evidence to support aggressive hypertension control, and availability of many new and effective antihypertensive drugs. It is clear that meaningful and sustained improvement in hypertension control will likely require fundamental changes in the current physician-centered office-visit based model of caring for hypertension. In this project we develop and implement an intervention that takes advantage of new technology and team models of care to improve BP measurement and control, solving the problems that have limited the application of case management approaches to hypertension care improvement. The study will take place in a diverse population of adults with hypertension cared for in a real-world primary care setting. The Telemonitoring Intervention (TI) integrates 2 innovative components: First, home BP measures are done using state-of-the-art modem-enabled automated equipment that internally stores and electronically transmits BP data through a simple touch-tone telephone connection to a secure web site. Second, a pharmacist case manager integrated with the primary care team through a jointly used electronic medical record (EMR) and formulary adjusts antihypertensive therapy using an approved written protocol, under a collaborative practice agreement with physicians. Treatment decisions are based on home BP data and are discussed and communicated to patients in telephone visits with the pharmacist case manager. Two-way communication between the pharmacist case manager and the patient's primary care team is assured by using a shared EMR and by additional secure messaging of the results of every pharmacist encounter to the primary care team. To assess the impact of the TI on hypertension control, patient satisfaction, and costs of care, we will conduct a cluster-randomized trial, assigning 16 primary care clinics and 450 of their nested patients with uncontrolled hypertension to either a Usual Care (UC) control group or TI. Blood pressure outcomes in both groups will be determined at baseline, 6, 12, 18 and 54 months in an identical and blinded fashion in a research clinic separate from the clinical setting where patients received their medical care. We hypothesize that guideline BP control will be achieved at 6 months and maintained at 12 months in more than 60% of patients from TI clinics, compared to < 40% in patients from UC clinics. We will compare satisfaction with care and costs in the TI and UC groups. The TI has the potential to improve hypertension control for millions of patients, and could be implemented widely in diverse and large patient populations based on performance in this randomized trial. The results of the project will have important implications for future efforts to improve care provided to many of the estimated 20 million Americans with uncontrolled hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or more
* Linked using EMR data to a HealthPartners Medical Group primary care clinic
* Within the 12-month period of time prior to screening have had at least 2 primary care outpatient encounters, in the two most recent of which the blood pressure was above Joint National Committee 7 (JNC7) goal (<140/90 mmHg or <130/80 for patients with diabetes or kidney disease).
* Have a measured blood pressure at a research clinic screening visit above the JNC7 goal

Exclusion Criteria:

* Acute coronary syndrome or stroke within the past 3 months
* Class III (marked limitation of physical activity) or IV (symptoms at rest) New York Heart Association heart failure, or known left ventricular ejection fraction (<30%)
* Severe renal dysfunction, with epidermal growth factor receptor (eGFR) ,30 ml/min/1.73 m2 using the abbreviated Modification of Diet in Renal Disease Study (MDRD) equation
* Known secondary causes of hypertension such as coarctation of the aorta, pheochromocytoma, adrenal cortical hypertension or renal vascular hypertension
* Unwillingness to be followed for a period of 18 months
* Pregnancy or unwillingness to use reliable bith control for females of child-bearing age
* Participation in another clinical trial
* Requires an interpreter to communicate with health care providers
* Dementia, mental illness or any condition that would limit ability to give informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2009-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Margolis, MD, MPH, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Margolis KL, Kerby TJ, Asche SE, Bergdall AR, Maciosek MV, O'Connor PJ, Sperl-Hillen JM. Design and rationale for Home Blood Pressure Telemonitoring and Case Management to Control Hypertension (HyperLink): a cluster randomized trial. Contemp Clin Trials. 2012 Jul;33(4):794-803. doi: 10.1016/j.cct.2012.03.014. Epub 2012 Apr 1. PMID 22498720
- [Background] Margolis KL, Asche SE, Bergdall AR, Dehmer SP, Maciosek MV, Nyboer RA, O'Connor PJ, Pawloski PA, Sperl-Hillen JM, Trower NK, Tucker AD, Green BB. A Successful Multifaceted Trial to Improve Hypertension Control in Primary Care: Why Did it Work? J Gen Intern Med. 2015 Nov;30(11):1665-72. doi: 10.1007/s11606-015-3355-x. PMID 25952653
- [Background] Pawloski PA, Asche SE, Trower NK, Bergdall AR, Dehmer SP, Maciosek MV, Nyboer RA, O'Connor PJ, Sperl-Hillen JM, Green BB, Margolis KL. A substudy evaluating treatment intensification on medication adherence among hypertensive patients receiving home blood pressure telemonitoring and pharmacist management. J Clin Pharm Ther. 2016 Oct;41(5):493-8. doi: 10.1111/jcpt.12414. Epub 2016 Jun 30. PMID 27363822
- [Background] Asche SE, O'Connor PJ, Dehmer SP, Green BB, Bergdall AR, Maciosek MV, Nyboer RA, Pawloski PA, Sperl-Hillen JM, Trower NK, Margolis KL. Patient characteristics associated with greater blood pressure control in a randomized trial of home blood pressure telemonitoring and pharmacist management. J Am Soc Hypertens. 2016 Nov;10(11):873-880. doi: 10.1016/j.jash.2016.09.004. Epub 2016 Sep 25. PMID 27720142
- [Result] Margolis KL, Asche SE, Bergdall AR, Dehmer SP, Groen SE, Kadrmas HM, Kerby TJ, Klotzle KJ, Maciosek MV, Michels RD, O'Connor PJ, Pritchard RA, Sekenski JL, Sperl-Hillen JM, Trower NK. Effect of home blood pressure telemonitoring and pharmacist management on blood pressure control: a cluster randomized clinical trial. JAMA. 2013 Jul 3;310(1):46-56. doi: 10.1001/jama.2013.6549. PMID 23821088
- [Result] Kerby TJ, Asche SE, Maciosek MV, O'Connor PJ, Sperl-Hillen JM, Margolis KL. Adherence to blood pressure telemonitoring in a cluster-randomized clinical trial. J Clin Hypertens (Greenwich). 2012 Oct;14(10):668-74. doi: 10.1111/j.1751-7176.2012.00685.x. Epub 2012 Jul 26. PMID 23031143
- [Derived] Margolis KL, Crain AL, Green BB, O'Connor PJ, Solberg LI, Beran M, Bergdall AR, Pawloski PA, Ziegenfuss JY, JaKa MM, Appana D, Sharma R, Kodet AJ, Trower NK, Rehrauer DJ, McKinney Z, Norton CK, Haugen P, Anderson JP, Crabtree BF, Norman SK, Sperl-Hillen JM. Comparison of explanatory and pragmatic design choices in a cluster-randomized hypertension trial: effects on enrollment, participant characteristics, and adherence. Trials. 2022 Aug 17;23(1):673. doi: 10.1186/s13063-022-06611-3. PMID 35978336
- [Derived] Margolis KL, Dehmer SP, Sperl-Hillen J, O'Connor PJ, Asche SE, Bergdall AR, Green BB, Nyboer RA, Pawloski PA, Trower NK, Maciosek MV. Cardiovascular Events and Costs With Home Blood Pressure Telemonitoring and Pharmacist Management for Uncontrolled Hypertension. Hypertension. 2020 Oct;76(4):1097-1103. doi: 10.1161/HYPERTENSIONAHA.120.15492. Epub 2020 Aug 31. PMID 32862713
- [Derived] Margolis KL, Asche SE, Dehmer SP, Bergdall AR, Green BB, Sperl-Hillen JM, Nyboer RA, Pawloski PA, Maciosek MV, Trower NK, O'Connor PJ. Long-term Outcomes of the Effects of Home Blood Pressure Telemonitoring and Pharmacist Management on Blood Pressure Among Adults With Uncontrolled Hypertension: Follow-up of a Cluster Randomized Clinical Trial. JAMA Netw Open. 2018 Sep 7;1(5):e181617. doi: 10.1001/jamanetworkopen.2018.1617. PMID 30646139
- [Derived] Annuzzi G, Bozzetto L, Costabile G, Giacco R, Mangione A, Anniballi G, Vitale M, Vetrani C, Cipriano P, Della Corte G, Pasanisi F, Riccardi G, Rivellese AA. Diets naturally rich in polyphenols improve fasting and postprandial dyslipidemia and reduce oxidative stress: a randomized controlled trial. Am J Clin Nutr. 2014 Mar;99(3):463-71. doi: 10.3945/ajcn.113.073445. Epub 2013 Dec 24. PMID 24368433

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was between March 2009-April 2011. We identified adult patients with elevated BP (systolic BP >140 or diastolic BP >90 mm Hg) at the two most recent primary care visits in the past year using electronic medical records. Patients received up to two mailings followed by phone calls. Further screening occurred in research clinic.
Pre-assignment Details: Participants were assigned to treatment group based on their primary care clinic location. Clinics were randomized to treatment or control (cluster randomization).
Groups:
- Telemonitoring Intervention: The telemonitoring intervention (TI) patients will receive a home blood pressure telemonitor and will work with a clinical pharmacist case manager to control elevated blood pressure. Patients will use their home telemonitors to read and send their blood pressures to their Pharmacist case manager, who will use phone meetings with the patient to make medication adjustments.
  Telemonitors and pharmacy management : Patients in the intervention arm will receive home blood pressure monitors, and will have individual hypertension case management from a medication therapy management pharmacist.
- Usual Care: Patients in the control group will receive usual care from their primary care physicians at HealthPartners Medical Group clinics.
Period: Overall Study
Arm/Group | Telemonitoring Intervention | Usual Care
Started | 228 | 222
Completed | 194 (completed both 6 and 12 month follow up) | 186 (completed both 6 and 12 month follow up)
Not Completed | 34 | 36
Not completed — Withdrawal by Subject | 13 | 8
Not completed — Did Not Attend Visit | 20 | 28
Not completed — Language barrier | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Telemonitoring Intervention | Total
Number analyzed (Participants) | 222 | 228 | 450
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 152 | 147 | 299
  >=65 years | 70 | 81 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (12.2) | 62.0 (11.7) | 61.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 103 | 201
  Male | 124 | 125 | 249
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 1 | 10
  Not Hispanic or Latino | 213 | 227 | 440
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 177 | 191 | 368
  Black or African American | 29 | 24 | 53
  Asian | 3 | 4 | 7
  Other | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Control
Description: Percentage of patients with controlled blood pressure at each time point (less than 140/90 mmHg or 130/80 mmHg for patients with kidney disease or diabetes)
Time Frame: Baseline, 6 months, 12 months, 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Usual Care | Telemonitoring Intervention
Number analyzed (Participants) | 222 | 228
percentage of participants
  Baseline | 0 [0 to 0] | 0 [0 to 0]
  6 Months | 45.2 [39.2 to 51.3] | 71.8 [65.6 to 77.3]
  12 Months | 52.8 [45.4 to 60.2] | 71.2 [62.0 to 78.9]
  18 Months | 57.1 [51.5 to 62.6] | 71.8 [65.0 to 77.8]

2. Primary Outcome: Mean Systolic Blood Pressure
Description: Systolic blood pressure at baseline and 4 time points
Time Frame: Baseline, 6 months, 12 months, 18 months, 54 months
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Usual Care | Telemonitoring Intervention
Number analyzed (Participants) | 222 | 228
mmHg
  Baseline | 147.7 [145.8 to 149.5] | 148.2 [146.3 to 150.0]
  6 Months | 136.9 [134.6 to 139.2] | 126.7 [124.4 to 129.0]
  12 Months | 134.8 [132.5 to 137.2] | 125.7 [123.4 to 128.0]
  18 Months | 133.0 [130.4 to 135.5] | 126.9 [124.3 to 129.4]
  54 Months | 131.7 [128.8 to 134.6] | 131.2 [128.3 to 134.1]

3. Primary Outcome: Mean Diastolic Blood Pressure
Description: Mean diastolic blood pressure at baseline and 4 time points
Time Frame: Baseline, 6 months, 12 months, 18 months, 54 months
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Usual Care | Telemonitoring Intervention
Number analyzed (Participants) | 222 | 228
mm Hg
  Baseline | 85.1 [82.9 to 87.3] | 84.4 [82.3 to 86.6]
  6 Months | 81.7 [79.5 to 84.0] | 75.0 [72.9 to 77.2]
  12 Months | 80.8 [78.5 to 83.2] | 75.1 [72.8 to 77.4]
  18 Months | 78.7 [76.6 to 80.9] | 75.1 [73.0 to 77.2]
  54 Months | 79.1 [76.8 to 81.4] | 77.8 [75.5 to 80.1]

ADVERSE EVENTS:
Time Frame: Events were reported at 6, 12, and 18 month clinic visits
Description: All events self-reported by participant
Arm/Group | Usual Care | Telemonitoring Intervention
Serious Adverse Events (participants affected / at risk) | 37/222 | 30/228
Other Adverse Events (participants affected / at risk) | 8/222 | 5/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Usual Care (N=222) | Telemonitoring Intervention (N=228)
Knee, hip, or shoulder arthroplasty (Surgical and medical procedures) | 2 (2) | 4 (4)
Acute pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 1 (3)
Spinal decompression/fusion (Surgical and medical procedures) | 6 (6) | 3/222 (3)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Worsening Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) — Secondary to other conditions (renal failure, Chronic Obstructive Pulmonary Disease(COPD ), GI blood loss, anal fissure)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Acute back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hashimoto's encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Fracture repair (Surgical and medical procedures) | 1 (1) | 2 (2) — Hospitalizations and surgery related to bone fracture
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Hernia repair (Surgical and medical procedures) | 1 (1) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Pyschiatric hospitalization (Psychiatric disorders) | 2 (2) | 1 (1) — Psychiatric hospital admissions: depression, alcohol abuse, psychosis, nonspecific altered mental state
Overdose, toxicity, or withdrawal (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) — Alcohol and narcotic overdose, toxicity, withdrawal
Prostate resection (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Peri-operative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0)
Hemorrhoid surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 2 (2) | 1 (1)
Bladder suspension (Surgical and medical procedures) | 1 (1) | 0 (0)
Ascites (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute abdominal pain (Hepatobiliary disorders) | 1 (1) | 0 (0) — Secondary to end stage liver disease
Chest pain, non-cardiac, non-specific (General disorders) | 4 (4) | 3 (4)
Chest pain, atypical (Cardiac disorders) | 0 (0) | 4 (4) — Cardiac cause not ruled out (history of cardiac disease, hypertensive crisis)
Hypertensive crisis (Cardiac disorders) | 1 (1) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (stroke) (Vascular disorders) | 5 (5) | 2 (2)
Hypotension with syncope (Vascular disorders) | 0 (0) | 3 (3) — Hospitalization for hypotension with syncope
Stable angina (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Transient Ischemic Attack (Vascular disorders) | 3 (3) | 0 (0)
Peripheral artery disease (Vascular disorders) | 1 (1) | 0 (0)
Coronary artery disease (Vascular disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 8 (8) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=222) | Telemonitoring Intervention (N=228)
Uretral stent change (Renal and urinary disorders) | 0 (0) | 1 (3)
Hypotension, dizziness, near syncope (Cardiac disorders) | 1 (1) | 3 (3) — ER or urgent care visit for low blood pressure, near syncope
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0) — ER or urgent care visit for high blood pressure
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) — New diagnosis
Allergic reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — ER visit for allergic reaction possibly related to antihypertensive drugs
Allergic vasculitis (Vascular disorders) | 1 (1) | 0 (0) — Secondary to bladder infection treatment

LIMITATIONS AND CAVEATS:
1) Response rate: 1 in 7 patients solicited by mail responded;of those screened, 1 in 4 eligible. 2) Participants were well-educated, had high income levels, 3) 1 integrated health care system, 4) study was not blinded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No